CLINICAL TRIAL: NCT03042299
Title: A Randomized, Open Label, 2-Period, 2-Treatment, Cross-over Phase 1 Study to Evaluate the Bio-equivalence of Single Oral Dose of TAK-536 Pediatric Formulation and TAK-536 Commercial Formulation in Healthy Adult Male Subjects
Brief Title: A Phase 1, Bio-equivalence Study of TAK-536 Pediatric Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Azilsartan-1004; U1111-1190-0845 (Registry Identifier: WHO); JapicCTI-173503 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Japanese Healthy Adult Male Participants
Keywords: Drug therapy
MeSH Terms: interventions — azilsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAK-536 Granules + TAK-536 Tablet (Experimental): TAK-536 10 milligram (mg), granules (pediatric formulation), under fasted condition, orally, once on Day 1 of Intervention Period 1, followed by a Washout Period of at least 6 days, further followed by TAK-536 10 mg, tablet (commercial formulation), under fasted condition, orally, once on Day 1 of Intervention Period 2.
  Interventions: Drug: TAK-536
- TAK-536 Tablet + TAK-536 Granules (Experimental): TAK-536 10 mg, tablet (commercial formulation), under fasted condition, orally, once on Day 1 of Intervention Period 1, followed by a Washout Period of at least 6 days, further followed by TAK-536 10 mg, granules (pediatric formulation), under fasted condition, orally, once on Day 1 of Intervention Period 2.
  Interventions: Drug: TAK-536

INTERVENTIONS:
Drug: TAK-536 — TAK-536 granules.
Drug: TAK-536 — TAK-536 tablet.

SUMMARY:
The purpose of this study is to evaluate the bio-equivalence of a single oral administration of TAK-536 pediatric formulation (granules) in comparison with a TAK-536 commercial formulation (tablet) in Japanese healthy adult male participants in an open label, 2-period, 2-treatment, cross-over design.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the bio-equivalence of a single oral administration of TAK-536 pediatric formulation (granules) in comparison with a TAK-536 commercial formulation (tablet) in healthy adult male participants in an open label, 2-period, 2-treatment, cross-over design.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator or sub-investigator, the participant is capable of understanding and complying with protocol requirements.
2. Signs and dates a written, informed consent form prior to the initiation of any study procedures.
3. Is a Japanese healthy adult male.
4. Aged 20 to 35 years, inclusive, at the time of informed consent.
5. Weighs at least 50.0 kilogram (kg), and has a body mass index (BMI) between 18.5 and 25.0 kilogram per square meter (kg/m^2), inclusive, at Screening.

Exclusion Criteria:

1. Has suspected hypotension with associated physical findings, such as dizziness postural, facial pallor, or cold sweats based on evaluation/physical examination at Screening, on the day before the study drug administration (Day -1) in Period 1, or up to the study drug administration on the Period 1.
2. Has received any study drug within 16 weeks (112 days) prior to the study drug administration in Period 1.
3. Has received TAK-536 or TAK-491 in a previous clinical study or as a therapeutic agent.
4. Has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
5. Has a known hypersensitivity to any component of the formulation of TAK-536 or any angiotensin II receptor blocker (ARB).
6. Has a positive urine drug result for drugs of abuse (defined as any illicit drug use) at Screening.
7. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 2 years prior to the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
8. Has taken any excluded medication, supplements, dietary products, or food products during the time periods specified in the protocol.
9. Has any current or recent (within 6 months) gastrointestinal diseases that would be expected to influence the absorption of drugs (that is, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [more than once per week] occurrence of heartburn, or any surgical intervention).
10. Has a history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Day 1 of Period 1.
11. Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody/antigen, or serological reactions for syphilis at Screening.
12. Has poor peripheral venous access.
13. Has undergone whole blood collection of at least 200 milliliter (mL) within 4 weeks (28 days) or at least 400 mL within 12 weeks (84 days) prior to the start of the study drug administration in Period 1.
14. Has undergone whole blood collection of at least 800 mL in total within 52 weeks (364 days) prior to the start of the study drug administration in Period 1.
15. Has undergone blood component collection within 2 weeks (14 days) prior to the start of the study drug administration in Period 1.
16. Has an abnormal (clinically significant) ECG at Screening or prior to the study drug administration in Period 1.
17. Has abnormal laboratory values that suggest a clinically significant underlying disease, or participant with the following laboratory abnormalities at Screening or prior to the study drug administration in Period 1: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) greater than (>) 1.5 * the upper limits of normal (ULN).
18. Who, in the opinion of the investigator or sub-investigator, is unlikely to comply with the protocol or is unsuitable for any other reason.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 14 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2017-03-11 (Actual); Study Completion 2017-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Nishi Kumamoto Hospital, Kumamoto, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 10 February 2017 to 11 March 2017.
Pre-assignment Details: Healthy male participants were enrolled in 1 of the 2 treatment sequences of this 2-period cross-over study to receive TAK-536 10 milligram (mg) granules (pediatric formulation) or TAK-536 10 mg tablet (commercial formulation).
Groups:
- TAK-536 Granules + TAK-536 Tablet: TAK-536 10 mg, granules (pediatric formulation), under fasted condition, orally, once on Day 1 of Intervention Period 1, followed by a Washout Period of at least 6 days, further followed by TAK-536 10 mg, tablet (commercial formulation), under fasted condition, orally, once on Day 1 of Intervention Period 2.
Period: Intervention Period 1 (6 Days)
Arm/Group | TAK-536 Granules + TAK-536 Tablet | TAK-536 Tablet + TAK-536 Granules
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Washout Period (at Least 6 Days)
Arm/Group | TAK-536 Granules + TAK-536 Tablet | TAK-536 Tablet + TAK-536 Granules
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Intervention Period 2 (6 Days)
Arm/Group | TAK-536 Granules + TAK-536 Tablet | TAK-536 Tablet + TAK-536 Granules
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-536 Granules + TAK-536 Tablet | TAK-536 Tablet + TAK-536 Granules | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.3 (0.95) | 21.3 (1.38) | 21.3 (1.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 7 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 7 | 7 | 14
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 167.7 (3.64) | 171.3 (4.42) | 169.5 (4.31)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 59.97 (5.586) | 60.49 (6.838) | 60.23 (6.005)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 21.33 (2.072) | 20.61 (2.143) | 20.97 (2.060)
Smoking classification [Count of Participants; unit: Participants]
  Never smoked | 5 | 4 | 9
  Current smoker | 1 | 3 | 4
  Ex-smoker | 1 | 0 | 1
Alcohol classification [Count of Participants; unit: Participants]
  Drank a few times per week | 1 | 2 | 3
  Drank a few times per month | 4 | 3 | 7
  Never drank | 2 | 2 | 4
Caffeine classification [Count of Participants; unit: Participants]
  Had caffeine consumption | 1 | 2 | 3
  Had no caffeine consumption | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-48): Area Under the Plasma Concentration-time Curve From Time 0 to 48 Hours Postdose for TAK-536
Time Frame: Day 1 pre-dose and at multiple time points post-dose (0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, and 48 hours post-dose; up to 48 hours)
Population: The pharmacokinetic (PK) analysis set included all participants who received the study drug, completed the minimum protocol-specified procedures without any major protocol deviations, and were evaluable for PK.
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Groups:
- TAK-536 10 mg Granules (Pediatric Formulation): TAK-536 10 mg, granules (pediatric formulation), under fasted condition, orally, once on Day 1 of either Intervention Period 1 or 2.
- TAK-536 10 mg Tablet (Commercial Formulation): TAK-536 10 mg, tablet (commercial formulation), under fasted condition, orally, once on Day 1 of either Intervention Period 1 or 2.
Arm/Group | TAK-536 10 mg Granules (Pediatric Formulation) | TAK-536 10 mg Tablet (Commercial Formulation)
Number analyzed (Participants) | 14 | 14
hour*nanogram per milliliter (h*ng/mL) | 6053.7 (1119.60) | 6479.6 (1008.00)
Statistical Analysis 1: Comparison: TAK-536 10 mg Granules (Pediatric Formulation) vs TAK-536 10 mg Tablet (Commercial Formulation); Test type: Equivalence — The difference in the least square (LS) means between formulations (TAK-536 pediatric formulation [granules]-TAK-536 commercial formulation [tablet]) and the two-sided 90 percent (%) confidence interval (CI) were provided using a crossover analysis of variance (ANOVA) model. The ANOVA model included log-transformed (natural log) PK parameters AUC 48 as dependent variable, and formulation, group, and period as independent variables; Point estimate = -0.0731, 90% CI 2-sided [-0.1088 to -0.0373]

2. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-536
Time Frame: as for outcome 1
Population: The PK analysis set included all participants who received the study drug, completed the minimum protocol-specified procedures without any major protocol deviations, and were evaluable for PK.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | TAK-536 10 mg Granules (Pediatric Formulation) | TAK-536 10 mg Tablet (Commercial Formulation)
Number analyzed (Participants) | 14 | 14
nanogram per milliliter (ng/mL) | 803.3 (113.63) | 878.1 (117.88)
Statistical Analysis 1: Comparison: TAK-536 10 mg Granules (Pediatric Formulation) vs TAK-536 10 mg Tablet (Commercial Formulation); Test type: Equivalence — The difference in the LS means between formulations (TAK-536 pediatric formulation [granules]-TAK-536 commercial formulation [tablet]) and the two-sided 90% CI were provided using a crossover ANOVA model. The ANOVA model included log-transformed (natural log) PK parameters Cmax as dependent variable, and formulation, group, and period as independent variables; Point estimate = -0.0909, 90% CI 2-sided [-0.1573 to -0.0244]

3. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-536
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | TAK-536 10 mg Granules (Pediatric Formulation) | TAK-536 10 mg Tablet (Commercial Formulation)
Number analyzed (Participants) | 14 | 14
h*ng/mL | 6187.4 (1167.72) | 6627.4 (1061.66)

4. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-536
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | TAK-536 10 mg Granules (Pediatric Formulation) | TAK-536 10 mg Tablet (Commercial Formulation)
Number analyzed (Participants) | 14 | 14
hours | 1.89 (0.738) | 2.43 (0.958)

5. Secondary Outcome: MRT∞,ev: Mean Residence Time After Extravascular Administration From Time 0 to Infinity for TAK-536
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | TAK-536 10 mg Granules (Pediatric Formulation) | TAK-536 10 mg Tablet (Commercial Formulation)
Number analyzed (Participants) | 14 | 14
hours | 9.781 (1.4010) | 10.11 (1.1873)

6. Secondary Outcome: Terminal Disposition Phase Rate Constant (λz) for TAK-536
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter per hour (L/h)
Arm/Group | TAK-536 10 mg Granules (Pediatric Formulation) | TAK-536 10 mg Tablet (Commercial Formulation)
Number analyzed (Participants) | 14 | 14
liter per hour (L/h) | 0.06866 (0.0046324) | 0.06862 (0.0077457)

7. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant who has signed informed consent to participate in a study; it does not necessarily have to have a causal relationship with this treatment or study participation. An AE can therefore be any unfavorable and unintended sign (for example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the study participation, whether or not it is considered related to the drug. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Baseline up to Day 6 of Intervention Period 2 (Day 18)
Population: The safety analysis set included all participants who received the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-536 10 mg Granules (Pediatric Formulation) | TAK-536 10 mg Tablet (Commercial Formulation)
Number analyzed (Participants) | 14 | 14
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With TEAEs Related to Vital Signs
Time Frame: Baseline up to Day 6 of Intervention Period 2 (Day 18)
Population: The safety analysis set included all the participants who received the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-536 10 mg Granules (Pediatric Formulation) | TAK-536 10 mg Tablet (Commercial Formulation)
Number analyzed (Participants) | 14 | 14
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With TEAEs Related to Body Weight
Time Frame: Baseline up to Day 6 of Intervention Period 2 (Day 18)
Population: The safety analysis set included all the participants who received the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-536 10 mg Granules (Pediatric Formulation) | TAK-536 10 mg Tablet (Commercial Formulation)
Number analyzed (Participants) | 14 | 14
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With TEAEs Related to Electrocardiograms (ECGs)
Time Frame: Baseline up to Day 6 of Intervention Period 2 (Day 18)
Population: The safety analysis set included all the participants who received the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-536 10 mg Granules (Pediatric Formulation) | TAK-536 10 mg Tablet (Commercial Formulation)
Number analyzed (Participants) | 14 | 14
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With TEAEs Related to Clinical Laboratory Tests
Time Frame: Baseline up to Day 6 of Intervention Period 2 (Day 18)
Population: The safety analysis set included all the participants who received the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-536 10 mg Granules (Pediatric Formulation) | TAK-536 10 mg Tablet (Commercial Formulation)
Number analyzed (Participants) | 14 | 14
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: TEAEs were assessed after the first dose of study drug until the follow up examination on Day 6 in Intervention Period 2 (Day 18)
Description: At each visit the investigator or sub-investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator or sub-investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-536 10 mg Granules (Pediatric Formulation) | TAK-536 10 mg Tablet (Commercial Formulation)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2016-12-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT03042299/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT03042299/SAP_001.pdf